CLINICAL TRIAL: NCT01194557
Title: Introducing Rapid Diagnostic Tests Into the Private Health Sector in Uganda: a Randomised Trial Among Registered Drug Shops to Evaluate Impact on Antimalarial Drug Use
Brief Title: Introducing Rapid Diagnostic Tests Into the Private Health Sector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: Ministry of Health, Uganda (Other Government); London School of Hygiene and Tropical Medicine (Other); Artemisinin-based Combination Therapy (Other)
Responsible Party: Principal Investigator, Pascal Magnussen, Senior Researcher, DBL -Institute for Health Research and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACTUGA3
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Fever; Malaria; Diagnosis; Referral
Keywords: history of fever; measured fever; appropriate treatment; appropriate referral
MeSH Terms: conditions — Fever; Malaria; Disease | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rapid diagnostic test (Active Comparator): Treatment and diagnosis of malaria in drugs hops using rapid diagnostic tests
  Interventions: Device: Rapid diagnostic test; Drug: Lumartem
- Presumptive malaria treatment (No Intervention): Presumptive treatment for malaria in drug shops

INTERVENTIONS:
Device: Rapid diagnostic test — Diagnosis of malaria using rapid diagnostic test
  Arms: rapid diagnostic test
Drug: Lumartem — Presumptive treatment of malaria/fever
  Arms: rapid diagnostic test

SUMMARY:
Most malaria deaths occur within 48 hours of onset of symptoms, and in rural areas with poor access to health facilities, home management of malaria (HMM) can improve the timeliness of treatment and reduce malaria mortality by up to 50%. In order to maximize both coverage and impact, artemisinin combination therapies (ACTs) should be deployed in HMM programmes, as well as in formal health facilities. Up to 80% of malaria cases are treated outside the formal health sector and shops are frequently visited as the first (and in some cases only) source of treatment. Strategies to deploy ACTs in Africa thus also need to examine the role of shops in home management and to ensure that drugs sold are appropriate. The current practice of presumptive treatment of any febrile illness as malaria (both at health facilities and in the context of HMM) based solely on clinical symptoms without routine laboratory confirmation, results in significant over-use of antimalarial drugs. With ACT being a more costly regimen, it is important to be more restrictive in its administration and rapid diagnostic tests (RDTs) provide a simple means of confirming malaria diagnosis in remote locations lacking electricity and qualified health staff.

This study therefore proposes to evaluate the feasibility, acceptability, and cost-effectiveness of using RDTs to improve malaria diagnosis and treatment by ocal drug shops in an area with high malaria transmission.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fever
* uncomplicted malaria

Exclusion Criteria:

* Complicated malaria
* known allergic reactions to Lumartem

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2600 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Appropriateness of treatment | 36 months

SECONDARY OUTCOMES:
Appropriateness of referral of complicated malaria cases | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony K Mbonye, PhD, Principal Investigator — Ministry of Health, Uganda
Locations (1):
- Mukono District, Mukono, Mukono, Uganda

REFERENCES:
- [Background] Chandler CI, Hall-Clifford R, Asaph T, Pascal M, Clarke S, Mbonye AK. Introducing malaria rapid diagnostic tests at registered drug shops in Uganda: limitations of diagnostic testing in the reality of diagnosis. Soc Sci Med. 2011 Mar;72(6):937-44. doi: 10.1016/j.socscimed.2011.01.009. Epub 2011 Feb 3. PMID 21349623
- [Background] Mbonye AK, Ndyomugyenyi R, Turinde A, Magnussen P, Clarke S, Chandler C. The feasibility of introducing rapid diagnostic tests for malaria in drug shops in Uganda. Malar J. 2010 Dec 21;9:367. doi: 10.1186/1475-2875-9-367. PMID 21176131
- [Derived] Hutchinson E, Hutchison C, Lal S, Hansen K, Kayendeke M, Nabirye C, Magnussen P, Clarke SE, Mbonye A, Chandler CIR. Introducing rapid tests for malaria into the retail sector: what are the unintended consequences? BMJ Glob Health. 2017 Jan 11;2(1):e000067. doi: 10.1136/bmjgh-2016-000067. eCollection 2017. PMID 28588992
- [Derived] Mbonye AK, Magnussen P, Lal S, Hansen KS, Cundill B, Chandler C, Clarke SE. A Cluster Randomised Trial Introducing Rapid Diagnostic Tests into Registered Drug Shops in Uganda: Impact on Appropriate Treatment of Malaria. PLoS One. 2015 Jul 22;10(7):e0129545. doi: 10.1371/journal.pone.0129545. eCollection 2015. PMID 26200467
- [Derived] Mbonye AK, Magnussen P, Chandler CI, Hansen KS, Lal S, Cundill B, Lynch CA, Clarke SE. Introducing rapid diagnostic tests for malaria into drug shops in Uganda: design and implementation of a cluster randomized trial. Trials. 2014 Jul 29;15:303. doi: 10.1186/1745-6215-15-303. PMID 25069975